CLINICAL TRIAL: NCT04432714
Title: A Phase II, Prospective, Single-center Study of Lenalidomide in Combination With R-DA-EPOCH in Patients With Untreated DLBCL With MYC Rearrangement
Brief Title: Lenalidomide in Combination With R-DA-EPOCH in Patients With Untreated DLBCL With MYC Rearrangement
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-430
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: DLBCL; Untreated; MYC Gene Rearrangement
Keywords: DLBCL; MYC Gene rearrangement; Lenalidomide; R-DA EPOCH
MeSH Terms: interventions — Lenalidomide; Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R2-DA-EPOCH (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 10mg/d#15mg/d#20mg/d#25mg/d d1~d10# 21days a cycle
Drug: Rituximab — Rituximab 375 mg/m2，IV, d0
Drug: Etoposide — Etoposide 50 mg/m2/day CI24h d1-d4
Drug: Doxorubicin — Doxorubicin 10 mg/m2/day CI24h d1-d4
Drug: Vincristine — Vincristine 0.4mg/m2/day CI24h d1-d4
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2/day IV d5
Drug: Prednisone — Prednisone 60 mg/m2/bid oral or IV d1-d5

SUMMARY:
The prognosis of DLBCL with MYC rearrangement is dismal. Previous study showed that lenalidomide in combination with R-CHOP showed promising therapeutic activity and that R-DA EPOCH was superior compared to R-CHOP regimen in this cohort of patients. The investigators therefore design this phase I/II study to investigate the safety and efficacy of lenalidomide in combination with R-DA EPOCH in patients with untreated MYC-rearranged DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL with MYC rearrangement according to WHO 2016 criteria, excluding PMBCL, PCNSL, HIV-associated lymphoma.
2. ECOG PS 0-2
3. Age 18-60 years old
4. Expected survival ≥ 12 weeks
5. A measurable or evaluable disease at the time of enrolment (diameter ≥1.5cm)
6. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Women who are pregnant or lactating. Patients have breeding intent in 12 months or cannot take effective contraceptive measures during the trial measures
2. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV infected persons
3. Previous exposure to any anti-tumor therapy
4. Poor hepatic and/or renal function, defined as total bilirubin, ALT, AST, Cr more than two fold of upper normal level,Ccr# 50 mL/min unless these abnormalities were related to the lymphoma
5. History of DVT or PE within past 12 months
6. Poor bone-marrow reserve, defined as neutrophil count less than 1.5×109/L or platelet count less than 75×109/L, unless caused by bone marrow infiltration
7. New York Heart Association class III or IV cardiac failure; or Ejection fraction less than 50%;or history of following disease in past 6 months: acute coronary syndrome#acute heart failure#severe ventricular arrhythmia
8. CNS or meningeal involvement
9. Known sensitivity or allergy to investigational product
10. Major surgery within three weeks
11. Patients receiving organ transplantation
12. Patients with secondary tumour, excluding cured (5 years without relapse) in situ Non-melanoma skin cancer. superficial bladder cancer, in situ cervical cancer, Gastrointestinal intramucous carcinoma and breast cancer
13. Presence of Grade III nervous toxicity within past two weeks
14. Active and severe infectious diseases
15. Any potential drug abuse, medical, psychological or social conditions whichmay disturb this investigation and assessment
16. In any conditions which investigator considered ineligible for this study
17. Patients with histological transformation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-06-09 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose and dose limited toxicity | 21 days after first cycle of R2-DA-EPOCH regimen (each cycle is 21 days)
Overall response rate | 6 months

SECONDARY OUTCOMES:
Progressive free survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Overall survival | 2 years
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Godfrey JK, Nabhan C, Karrison T, Kline JP, Cohen KS, Bishop MR, Stadler WM, Karmali R, Venugopal P, Rapoport AP, Smith SM. Phase 1 study of lenalidomide plus dose-adjusted EPOCH-R in patients with aggressive B-cell lymphomas with deregulated MYC and BCL2. Cancer. 2019 Jun 1;125(11):1830-1836. doi: 10.1002/cncr.31877. Epub 2019 Feb 1. PMID 30707764
- [Background] Coiffier B, Sarkozy C. Diffuse large B-cell lymphoma: R-CHOP failure-what to do? Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):366-378. doi: 10.1182/asheducation-2016.1.366. PMID 27913503
- [Background] Dunleavy K, Fanale MA, Abramson JS, Noy A, Caimi PF, Pittaluga S, Parekh S, Lacasce A, Hayslip JW, Jagadeesh D, Nagpal S, Lechowicz MJ, Gaur R, Lucas A, Melani C, Roschewski M, Steinberg SM, Jaffe ES, Kahl B, Friedberg JW, Little RF, Bartlett NL, Wilson WH. Dose-adjusted EPOCH-R (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab) in untreated aggressive diffuse large B-cell lymphoma with MYC rearrangement: a prospective, multicentre, single-arm phase 2 study. Lancet Haematol. 2018 Dec;5(12):e609-e617. doi: 10.1016/S2352-3026(18)30177-7. PMID 30501868